CLINICAL TRIAL: NCT02568839
Title: PREDIX HER2 - Neoadjuvant Response-guided Treatment of HER2 Positive Breast Cancer. Part of a Platform of Translational Phase II Trials Based on Molecular Subtypes
Brief Title: Neoadjuvant Response-guided Treatment of HER2 Positive Breast Cancer
Acronym: PREDIX HER2
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Thomas Hatschek (Other)
Responsible Party: Sponsor-Investigator, Thomas Hatschek, Sen. Consultant, MD, PhD, Assoc. professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREDIX HER2
Record Dates: First submitted 2015-09-21; First posted 2015-10-06 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Early-Stage Breast Carcinoma; HER-2 Positive Breast Cancer
Keywords: Neoadjuvant therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; pertuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A standard treatment (Active Comparator): docetaxel + trastuzumab sc + pertuzumab. Treatment with all three drugs is given on day 1, repeated every three weeks. Six courses of preoperative treatment. Response evaluations after every 2nd course. In case of no change (NC), treatment is switched to arm B.
  Postoperatively, patients receive 2 courses of treatment with the combination epirubicin + cyclophosphamide (EC), followed by adjuvant trastuzumab, radiotherapy, eventually endocrine treatment.
  Interventions: Drug: docetaxel + trastuzumab sc + pertuzumab
- B experimental treatment (Experimental): trastuzumab emtansine. Treatment is given on day 1, repeated every three weeks. Six courses of preoperative treatment. Response evaluations after every 2nd course. In case of no change (NC), treatment is switched to arm A.
  Postoperatively, patients receive 4 courses of treatment with the combination epirubicin + cyclophosphamide (EC), followed by adjuvant trastuzumab, radiotherapy, eventually endocrine treatment.
  Interventions: Drug: trastuzumab emtansin

INTERVENTIONS:
Drug: docetaxel + trastuzumab sc + pertuzumab — docetaxel 75-100 mg IV + trastuzumab sc 5 ml (600 mg) SC + pertuzumab 840 mg IV starting dose, subsequently 420 mg IV, repeated every 3 weeks, 6 courses
  Other Names: Herceptin SC; Perjeta
  Arms: A standard treatment
Drug: trastuzumab emtansin — trastuzumab emtansine 3.6 mg/kg IV, repeated every 3 weeks, 6 courses
  Other Names: Kadcyla
  Arms: B experimental treatment

SUMMARY:
The purpose of this trial is to evaluate efficacy and toxicity of either the combination of docetaxel, trastuzumab sc and pertuzumab (arm A) or trastuzumab emtansin (arm B). Switch of therapy to the opposite treatment alternative is applicable in case of lack of response after two courses of treatment, or for medical reasons under exceptional circumstances (drug reaction, other medical conditions) at any point. After termination of the primary treatment follow-up for five years.

A translational subprotocol is a mandatory part of the study protocol, with exception for the use of PET-CT evaluations.

DETAILED DESCRIPTION:
Patients with HER2-positive tumors >20 mm or verfied regional lymph node metastases are randomized to either arm A, the combination of docetaxel, trastuzumab sc (Herceptin SC®) and pertuzumab (Perjeta®) or arm B, trastuzumab emtansin (Kadcyla®). Switch to the opposite treatment is performed in case of lack of response after evaluations with mammography and ultrasound, alternatively MRI breast after the 2nd, 4th and 6th course of treatment.

Postoperative treatment, trastuzumab, radiotherapy, eventual endocrine treatment) according to standard guidelines. Structured follow-up visits yearly for five years, including reporting of persistent treatment-related toxicity, HRQoL, recurrence and death.

The trial contains also a translational subprotocol:

1. PET-CT using FDG, confined to the chest, is performed before start, and after the 2nd and 6th course (functional imaging, optional).
2. Core biopsies from the tumor are collected before start and after the 2nd course of treatment. If residual tissue is available, samples are collected from the surgical sample
3. Blood samples are collected repeatedly during the ongoing treatment and yearly follow-up
4. FNAs from metastases in case of recurrence during follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Patients with breast cancer confirmed by histology, characterized by immunohistochemistry for ER, PR, HER2 and proliferation marker
3. Tumor and blood samples available. HER2 type confirmed by ISH
4. Age 18 years or older. Elderly patients in condition adequate for planned therapy
5. Primary breast cancer >20mm in diameter and/or verified lymph node metastases
6. Adequate bone marrow, renal, hepatic and cardiac functions and no other uncontrolled medical or psychiatric disorders
7. LVEF ≥55%
8. ECOG performance status 0-1
9. Primary breast cancer as defined in p. 5 plus at most 2 morphologically characterized well-defined distant metastases accessible for stereotactic radiotherapy, provided that this treatment is available

Exclusion Criteria:

1. Distant metastases, including node metastases in the contralateral thoracic region or in the mediastinum
2. Other malignancy diagnosed within the last five years, except for radically treated basal or squamous cell carcinoma of the skin or CIS of the cervix
3. Patients in child-bearing age without adequate contraception
4. Pregnancy or lactation
5. Uncontrolled hypertension, heart, liver, kidney related or other medical or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2014-11; Primary Completion 2019-02 (Actual); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Pathological objective response to primary medical treatment | At surgery
  Efficacy measure after 18 weeks of preoperative treatment, starting from the start of preoperative medical treatment until the date of surgery. Outcome should be received within not more than 4 weeks post surgery

SECONDARY OUTCOMES:
Clinical/radiological objective response during neoadjuvant treatment | During the 18-week treatment period before surgery
  Clinical measurements with caliper, radiological evaluations with mammography and ultrasound, alternately MRI, within 6 weeks before start, and 14 days after 3-weekly courses 2, 4 and 6; PET-CT within 2 weeks before start, and 16 days after courses 2 and 6. Time frame for these response evaluations is between between week 4 and week 18 of preoperative treatment
Event-free survival | All events from date of randomization until follow-up to 10 years
  Time frame for reporting is from date of randomization until first reported event, including disease progression, documented first recurrence, first contralateral breast cancer, first cancer of other origin, or death of any cause, whatever occurs first
Disease-free survival | During the follow-up to 10 years
  Time frame for reporting is between date of surgery and 10 years follow-up. Date of detection of metastasis will be reported within 12 months after occurence
Breast cancer specific survival | During the follow-up to 10 years
  Time frame for reporting is between date of surgery and 60 months follow-up. Date and cause of death will be reported within 12 months after occurence
Overall survival | During the follow-up to 10 years
  Time frame for reporting is between date of surgery and 10 years follow-up. Date of death will be reported within 12 months after occurence
Incidence of treatment-emergent adverse events [Safety and Tolerability] | During the 18-week period of treatment and until 30 days after termination and during the follow-up period up to 10 years
  Time frame for reporting of acute side effects is from start of treatment until 30 days after termination of the treatment, totally 22 weeks. Late side effects are reported within 60 months post surgery. Cardiac toxicity is given special attention during the entire period. Echocardiograms and ECGs are performed within 6 weeks before start of treatment, after 16 weeks of treatment before surgery, and then every 3 months during postoperative treatment with trastuzumab the 1st postoperative year; thereafter every 12 months until 10 years of follow-up after surgery
Health Related Quality of life | From date of randomisation until follow-up to 5 years
  Repeated assessments using EOTC QLQ-C30 and BR23 during the treatment period, before randomization and after courses 2, 4 and 6, 3 months post surgery and annually during the follow-up period up to 10 years. Time frame covers the 18-week period of preoperative treatment and 10 years follow-up period after surgery
Frequency of breast-conserving surgery | At surgery
  Type of surgery is recorded at the time of surgery

OTHER OUTCOMES:
Changes of morphological, functional and biological characteristics of early breast cancer before and after exposure to cytotoxic and targeted treatment | 5 years
  Includes genomics, proteomics and other biomarker-related analyses on core biopsies and blood samples before start and after two courses of treatment, collection of tumor samples from the surgical specimen at the date of operation, blood samples in connection with annual follow-up visits and FNA and blood samples in case of recurrence. Time frame for collection of biological samples from start of preoperative treatment until 60 months of follow-up post surgery. Functional imaging using 18F-FDG PET-CT is performed at baseline and after the 2nd and 6th treatment course.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hatschek, Assoc prof, Study Chair — Breast-sarcoma unit, Dept. of Oncology, Karolinska university hospital; Jonas Bergh, Professor, Study Director — Dept. of Oncology-Pathology, Karolinska Institutet
Locations (7):
- Sweden (7):
  - Dept. of Oncology, Örebro University Hospital, Örebro, Närke
  - Dept. of Oncology, Sahlgrenska University Hospital, Gothenburg
  - Dept. of Oncology, Skåne University Hospital, Lund
  - Dept. of Oncology, Karolinska University Hospital, Stockholm
  - Dept. of Oncology, Sundsvall Hospital, Sundsvall
  - Dept. of Oncology, University Hospital of Umeå, Umeå
  - Dept. of Oncology, Uppsala University Hospital, Uppsala

REFERENCES:
- [Derived] Zhu Y, Zerdes I, Matikas A, Cruz IR, Bergqvist M, Elinder E, Bosch A, Lindman H, Einbeigi Z, Andersson A, Carlsson L, Dreifaldt AC, Isaksson-Friman E, Hellstrom M, Johansson H, Wang K, Bergh JCS, Hatschek T, Foukakis T. The role of serum thymidine kinase 1 activity in neoadjuvant-treated HER2-positive breast cancer: biomarker analysis from the Swedish phase II randomized PREDIX HER2 trial. Breast Cancer Res Treat. 2024 Apr;204(2):299-308. doi: 10.1007/s10549-023-07200-x. Epub 2024 Jan 4. PMID 38175448
- [Derived] Matikas A, Johansson H, Gryback P, Bjohle J, Acs B, Boyaci C, Lekberg T, Fredholm H, Elinder E, Margolin S, Isaksson-Friman E, Bosch A, Lindman H, Adra J, Andersson A, Agartz S, Hellstrom M, Zerdes I, Hartman J, Bergh J, Hatschek T, Foukakis T. Survival Outcomes, Digital TILs, and On-treatment PET/CT During Neoadjuvant Therapy for HER2-positive Breast Cancer: Results from the Randomized PREDIX HER2 Trial. Clin Cancer Res. 2023 Feb 1;29(3):532-540. doi: 10.1158/1078-0432.CCR-22-2829. PMID 36449695
- [Derived] Hatschek T, Foukakis T, Bjohle J, Lekberg T, Fredholm H, Elinder E, Bosch A, Pekar G, Lindman H, Schiza A, Einbeigi Z, Adra J, Andersson A, Carlsson L, Dreifaldt AC, Isaksson-Friman E, Agartz S, Azavedo E, Gryback P, Hellstrom M, Johansson H, Maes C, Zerdes I, Hartman J, Brandberg Y, Bergh J. Neoadjuvant Trastuzumab, Pertuzumab, and Docetaxel vs Trastuzumab Emtansine in Patients With ERBB2-Positive Breast Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 Sep 1;7(9):1360-1367. doi: 10.1001/jamaoncol.2021.1932. PMID 34165503
- See also: Oral presentation, #97O, at ESMO Breast conference 2020. — http://esmo.org